CLINICAL TRIAL: NCT00845377
Title: Changing Minds - Studying the Effects of a Tailored Psychosocial Support Model on Depressive Mood and Quality of Life in Depressive Elderly People
Brief Title: Changing Minds - Supporting Depressed Elderly People With an Individually Tailored Service Model
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Union for the Welfare of the Aged (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Marja Saarenheimo, Senior researcher, Central Union for the Welfare of the Aged
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUWAged 0901
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Depression; Psychological Well-Being
Keywords: Depression; Aging; Psychological well-being; Psychosocial intervention
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Counseling (Experimental)
  Interventions: Behavioral: Comprehensive psychosocial support for depressed elderly

INTERVENTIONS:
Behavioral: Comprehensive psychosocial support for depressed elderly — The model includes a psychiatric nurse as a care manager, a multiprofessional team with a physiotherapist, psychologist and psychiatrist. Each participant receives individually tailored services such as therapeutic groups, conversation groups, physical exercise, music therapy, art therapy and nutritional counseling
  Other Names: Supporting elderly people with depression; Mental health counseling for elderly people; Individually tailored support model for old age depression

SUMMARY:
Depression is one of the leading causes of emotional suffering in later life. It has been estimated that 2-5% of community-dwelling elderly people suffer from major depression, but according to recent studies, as much as 25 % have clinically significant depressive symptoms.Typically, depressive symptoms in the elderly are treated solely with antidepressants.

The aim of this project is to study the effects of a comprehensive psychosocial intervention on the psychological well-being, quality of life and use of services in depressed elderly people. In addition, the processes of intervention are studied from the perspective of the participants as well as the service system. The research is conducted in collaboration with the city of Espoo. The design of the study combines clinical trial with qualitative process analysis.

ELIGIBILITY:
Inclusion Criteria:

* age 60+

Exclusion Criteria:

* severe memory disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Alleviating depressive symptoms measured with Geriatric Depression Scale | base line, 6 months, 1 year

SECONDARY OUTCOMES:
Quality of life measured with WHO QuolBref | base line, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marja K Saarenheimo, PhD, Study Director — Central Union for the Welfare of the Aged
Locations (1):
- Central Union for the Welfare of the Aged, Helsinki, Finland